CLINICAL TRIAL: NCT03505554
Title: A Phase 2 Open Label Study of Oral Lorlatinib in Patients With Relapsed ALK Positive Lymphoma Previously Treated With ALK Inhibitors (CRU3)
Brief Title: A Study of Oral Lorlatinib in Patients With Relapsed ALK Positive Lymphoma
Acronym: CRU3
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milano Bicocca (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRU3
Record Dates: First submitted 2018-04-06; First posted 2018-04-23 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Anaplastic Large Cell Lymphoma, ALK-Positive
Keywords: ALK; relapsed; lorlatinib
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Recurrence | interventions — lorlatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lorlatinib (Experimental): 100 mg QD
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — 100 mg QD
  Other Names: PF-06463922

SUMMARY:
The purpose of this study is to define the objective response rates (ORR) of Lorlatinib in subjects with ALK+ lymphomas resistant or refractory to ALK inhibitors.

DETAILED DESCRIPTION:
Lorlatinib is a selective and potent tyrosine kinase inhibitor of ALK and ROS1 that pre-clinically demonstrated dose-dependent inhibition of mutations that confer resistance to other ALK inhibitors; it is also a brain-penetrant thus it might be active in patients with CNS metastases.

Study Objectives Primary Define the objective response rates (ORR) of PF-06463922 in subjects with ALK+ lymphomas resistant or refractory to ALK inhibitors.

Secondary

* Define the Progression Free Survival (PFS) in subjects with ALK+ lymphomas resistant or refractory to ALK inhibitors.
* Define the overall survival (OS) in ALK+ lymphoma patients treated with Lorlatinib, that are resistant or refractory to ALK inhibitors.
* Determine the toxicity profile of Lorlatinib in ALK+ lymphoma patients resistant or refractory to ALK inhibitors.
* Determine the Quality of Life (QoL) in this population of patients using the EORTC-C30 Quality of Life questionnaire.
* Study the mutational status of ALK pre/post Lorlatinib treatment through next-generation sequencing (NGS).

Study design This is a phase 2 study open to 12 eligible patients with lymphoma with a confirmed ALK rearrangement. All patients must have been pretreated with at least one line of standard cytotoxic chemotherapy and at least one ALK inhibitor and they must have demonstrated progression (regardless of initial response) or resistance on the last treatment.

The study begins with a screening period to assess eligibility, up to and including 28 days prior to the first dose of Lorlatinib. Treatment will continue until patient experiences unacceptable toxicity or progressive disease (PD), starts a new anti-cancer therapy or dies.

The study will remain open until all patients have completed 3 years from the enrollment.

Study treatment Patients will receive an oral administration of Lorlatinib at a dose of 100mg QD. In case of toxicity, it is possible to proceed to a dose reduction (75mg or 50mg QD) or a temporary interruption of Lorlatinib.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated Informed Consent approved by Local Ethical Committee before any protocol-specific screening procedures.
2. ALK+ Lymphoma diagnosed by IHC or FISH.
3. Refractory disease or relapse after at least one prior chemotherapy regimen (typically a minimum of 6 cycles of CHOP) and at least one ALK inhibitor; presence of measurable disease by physical examination, CT or CT-PET scan.
4. Any prior antitumor medical treatment or major surgeries must have been completed at least 14 days prior to initiation of study medication. This could not be respected if there is clear evidence of disease progression, manifested as growing pain attributable to the tumour, fever, growing tumour lesions, increasing LDH values. Systemic anti-cancer therapy completed within a minimum of 5 half-lives of study entry.
5. Able to take oral therapy.
6. Female or male, 18 years of age or older.
7. ECOG performance status 0-3.
8. Adequate organ function as defined by the following criteria:

   Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤ 2.5 x upper limit of normal (ULN) or AST and ALT ≤ 5 x ULN if liver function abnormalities are due to underlying malignancy Total serum bilirubin 1.5 x ULN (except patients with documented Gilbert's syndrome Creatinine ≤ 1.5 x ULN.
9. Adequate bone marrow function:

   Absolute neutrophil count (ANC) ≥ 1000/µL Platelets ≥ 50.000/µL Hemoglobin ≥ 9.0 g/dL The hematological values will not be considered in case of bone marrow involvement.
10. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
11. Female and male patients who are of childbearing potential must agree to use an effective form of contraception (2 forms of contraception) with their partners throughout participation in this study and for at least 90 days after the last dose of treatment.

Exclusion Criteria:

1. Current treatment on another therapeutic clinical trial.
2. Clinically significant cardiovascular disease (that is, active or <3 months prior to enrollment): cerebral vascular accident/stroke, myocardial infarction, unstable angina, congestive heart failure (New York Heart Association Classification Class ≥ II)
3. Ongoing cardiac dysrhythmias of NCI CTCAE Grade ≥2: second-degree or third-degree AV block (unless paced) or any AV block with PR >220 msec, uncontrolled atrial fibrillation of any grade, bradycardia defined as <50 bpm (unless patient is otherwise healthy such as long-distance runners, etc.), machine-read ECG with QTc >470 msec, or congenital long QT syndrome.
4. Pregnancy or breastfeeding.
5. Use of drugs or foods that are known strong or moderate CYP3A4 inhibitors, inducers and substrates; drugs that are CYP2C9 substrates; drugs that are strong CYP2C19 inhibitors; drugs that are strong CYP2C8 inhibitors; and drugs that are P-gp substrates.
6. Prior malignancy other than basal cell carcinoma , if original diagnosis happened in the last 5 years.
7. Patients with predisposing characteristics for acute pancreatitis according to investigator judgment (e.g. uncontrolled hyperglycemia, current gallstone disease, alcoholism).
8. Hypertriglyceridemia ≥ grade 1.
9. Active and clinically significant bacterial, fungal, or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS) related illness.
10. Other severe acute or chronic medical or psychiatric conditions, or laboratory abnormalities that would impart, in the judgment of the investigator and/or sponsor, excess risk associated with study participation or study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-10-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 1 year
  ORR

SECONDARY OUTCOMES:
Progression Free Survival | 1 year
  PFS
Overall Survival | 1 year
  OS
toxicity | up to 24 months
  number, type and grade of adverse events
Quality of life | up to 24 months
  Use of EORTC-QLQ-C30 questionnaire
Study the mutational status of ALK pre/post Lorlatinib | up to 24 months
  Mutational Analysis

CONTACTS AND LOCATIONS:
Overall Officials: CARLO GAMBACORTI-PASSERINI, MD, Principal Investigator — University of Milano Bicocca
Locations (2):
- Italy (2):
  - Asst-Monza, Monza, Italy/MB
  - UOC Ematologia, Ospedale S. Eugenio, Roma